CLINICAL TRIAL: NCT05308576
Title: A Randomized, Double-blind, Parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of SCTV01E (Alpha/Beta/Delta/Omicron Variants S-Trimer COVID-19 Vaccine) in Population Aged ≥18 Years
Brief Title: A Study to Evaluate the Efficacy and Safety of SCTV01E (a COVID-19 Vaccine) in Population Aged ≥18 Years
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCTV01E-MRCT-2
Record Dates: First submitted 2022-02-11; First posted 2022-04-04 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 infection; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTV01E (Experimental): one dose of SCTV01E on D0
  Interventions: Biological: SCTV01E
- Placebo (Placebo Comparator): one dose of Placebo on D0
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SCTV01E — D0; intramuscular injection
  Arms: SCTV01E
Biological: Placebo — D0; intramuscular injection
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effectiveness of SCTV01E in participants aged ≥18 years.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled Phase III study. It will evaluate the protective effectiveness and safety of SCTV01E against COVID-19 in participants who were previously received primary series or booster dose of COVID-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years old when signing ICF;
2. Participants who were fully vaccinated with COVID-19 vaccine and/or received booster vaccination, and the interval between the last dose of COVID-19 vaccine previously received and screening is 6 to 24 months;
3. The participant and/or his/her legal representative can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. The participant and/or his/her legal representative have the ability to read, understand, and fill in record cards;
5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, Chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
6. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the last dose of study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

1. A positive result of nucleic acid test or rapid antigen test for SARS-CoV-2 during the screening period;
2. Presence of fever within 3 days before the study vaccination;
3. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
4. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
5. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
6. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
7. Patients on antituberculosis therapy;
8. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (skin basal cell carcinoma and carcinoma in-situ of cervix are exceptions and will not be excluded), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
9. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
10. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
11. Participants who received other investigational drugs within 1 month before the study vaccination;
12. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
13. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
14. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
15. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
16. Those who plan to donate ovum or sperms during the study period;
17. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
18. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
19. Those who are tested positive for HIV in terms of serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Cases of the first occurrence of symptomatic COVID-19 of any severity starting 7 days (≥8 days) after the study vaccination | 7 days after the study vaccination
  After the study vaccination, participants were contacted weekly to inquire about any signs or symptoms related to COVID-19. Participants were encouraged to report any COVID-19-related symptoms they experienced spontaneously during the study period.

SECONDARY OUTCOMES:
cases of the first occurrence of all infection, asymptomatic infection, infection with multiple symptoms, moderate, severe, and death due to COVID-19, starting 7-days post-vaccination | 7 days after the study vaccination
  Participants were contacted weekly to inquire about any signs or symptoms related to COVID-19. Participants were encouraged to report any COVID-19-related symptoms they experienced spontaneously during the study period.
Cases of the first occurrence of all infection, asymptomatic infection, symptomatic infection, infection with multiple symptoms, respectively, starting 14-days post- vaccination. | 14 days after the study vaccination
  Participants were contacted weekly to inquire about any signs or symptoms related to COVID-19. Participants were encouraged to report any COVID-19-related symptoms they experienced spontaneously during the study period.
Cases of the first occurrence of symptomatic infection, infection with multiple symptoms, moderate, severe and death due to COVID-19, caused by SARS-CoV-2 variants, starting 14-days post-vaccination. | 14 days after the study vaccination
  Participants were contacted weekly to inquire about any signs or symptoms related to COVID-19. Participants were encouraged to report any COVID-19-related symptoms they experienced spontaneously during the study period.
Immunogenicity: GMT of neutralizing antibody (nAb) against SARS-CoV-2 variants or subvariants on 7, 14, 28, 90, 180 and 365 days post-vaccination | Day 0, Day 7, Day 14, Day 28, Day 90, Day 180 and Day 365
  Blood samples were collected from participants in the immunogenicity subgroup on 0 (pre-injection), 14, and 28 days post-vaccination. Additional blood samples were collected from 200 participants in the immunogenicity subgroup on 7, 90, 180 and 365 days post-vaccination for geometric mean titers (GMTs) of live virus neutralizing antibodies against Omicron BA.5 variant using 50% plaque reduction neutralization test (PRNT50).
Immunogenicity: Seroresponse rate of nAb against SARS-CoV-2 (including its variants and subvariants) on Day 7, Day 14, Day 28, Day 90, Day 180 and Day 365. | Day 0, Day 7, Day 14, Day 28, Day 90, Day 180 and Day 365
  the sereresponse rates (SRRs) of nAb (change from <lower limit of quantification (LLOQ) to ≥4 ×LLOQ, or at least a fourfold rise if baseline ≥LLOQ) compared with the pre-injection baseline (95%CI) against SARS-CoV-2 variants or subvariants
Safety: Incidence and severity of solicited AEs of SCTV01E from D0 to D7. | Day 0 to Day 7 after the study vaccination.
  Both active monitoring and spontaneous reporting were used. Solicited AEs within 7 days after the study vaccination were collected through vaccination record cards (VRCs).
Safety: Incidence and severity of unsolicited AEs of SCTV01E from D0 to D28. | Day 0 to Day 28 after the study vaccination.
  Both active monitoring and spontaneous reporting were used. Unsolicited AEs within 28 days after the study vaccination were collected through vaccination record cards (VRCs).
Safety: Incidence and severity of SAEs and AESIs from D0 to D365. | Day 0 to Day 365 after the study vaccination.
  Serious adverse events (SAEs) and adverse events of special interest (AESIs) were collected by investigators via phone calls, short messages, e-mails, visits on-site, or other contact methods for up to 365 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Guizhou center for disease control and prevention, Guiyang, Guizhou, China

REFERENCES:
- [Derived] Yan L, Yi J, Liu D, Li J, Baidoo AAH, Xie L. Baseline Anti-SARS-CoV-2 IgG and Protection from Symptomatic Infection: Post Hoc Analysis of the SCTV01E Phase 3 Randomized Trial. Vaccines (Basel). 2025 Sep 19;13(9):984. doi: 10.3390/vaccines13090984. PMID 41012186